CLINICAL TRIAL: NCT00128856
Title: Phase II Pharmacogenomic and Clinical Trial for the Administration of Gemcitabine-doxorubicin-paclitaxel (GAT) as Neoadjuvant Treatment of Patients With Stage III Breast Cancer
Brief Title: Gemcitabine, Doxorubicin and Paclitaxel (GAT) as Neoadjuvant Treatment of Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Eli Lilly and Company (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM 2002-01
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant chemotherapy.; Stage III disease.
MeSH Terms: conditions — Breast Neoplasms; Disease | interventions — Gemcitabine; Doxorubicin; Paclitaxel

ARMS (1):
- Gemcitabine + Adriamycine + Paclitaxel (Experimental): Neoadjuvant chemotherapy consisted of adriamycine 40 mg/m2, administered on day 1 as an i.v. infusion. Paclitaxel 150 mg/m2 was administered on day 2 as an i.v infusion followed by gemcitabine 2000 mg/m2 as an i.v. infusion. The three drugs were administered every two weeks for 6 cycles.
  Interventions: Drug: Gemcitabine; Drug: Adriamycine; Drug: Paclitaxel

INTERVENTIONS:
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Adriamycine
  Other Names: doxorubicin
Drug: Paclitaxel
  Other Names: Taxol

SUMMARY:
This is a multicenter, open-label, phase II trial to assess the efficacy of the GAT neoadjuvant regimen in patients with stage III breast cancer.

DETAILED DESCRIPTION:
2 treatment cycles of chemotherapy (one cycle = 2 weeks) must be administered to each patient before breast surgery.

The required number of patients has been calculated following Simon's method. 43 patients will be enrolled in two phases: first, 29 patients must be enrolled, and at least 2 pathological complete responses obtained. Patients recruitment will continue until 43 patients have been enrolled. Assumptions are that there is a 95% probability to obtain a rate of pathological complete responses of at least 10%.

ELIGIBILITY:
Inclusion Criteria:

* Stage III breast cancer disease, with histological confirmation by true-cut or open-biopsy.
* Ages between 18 and 75 years old. Patients older than 70 must have an adequate quality of life to be eligible.
* Patients cannot have received previous treatment with chemotherapy, hormone therapy, radiotherapy or immune therapy.
* Performance status of 0,1, 2 Eastern Cooperative Oncology Group (ECOG).
* At least a 6 month life expectancy.
* Neutrophils > 1500; platelets > 100000; haemoglobin > 10 mg/dL.
* Adequate renal and hepatic functions, with serum creatinine < 1.2 mg/dl and total bilirubin < 2 mg/dl.
* Adequate contraceptive methods during the study and up to 3 months after.
* Adequate cardiac function assessed by physical exam, electrocardiogram and left ventricular ejection fraction > 55%.

Exclusion Criteria:

* Inflammatory carcinoma or stage I, II or IV breast cancer disease.
* Males.
* Active infection.
* Other neoplasms except for basal skin carcinoma or cervical in situ carcinoma adequately treated. Other previous neoplasms are allowed if diagnosed and treated more than 5 years before study registration.
* Concomitant serious disease provoking organ failure (heart, renal, hepatic, respiratory).
* Pre-existing motor or sensorial neuropathy > grade 1.
* Inability for treatment compliance.
* History of hypersensitivity to compounds such as cremophor, cyclosporine or vitamin K.
* History of arrhythmias or congestive heart failure, even when controlled; or active cardiac blocking of second or third grade.
* History of myocardial infarction in the previous 6 months.
* Hypertension not controlled.
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-03 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Up to week 15
  pCR is defined as no invasive cells identifiable in breast sections at surgery. Response will be measured by physical exam and breast imaging before surgery and will be evaluated according to the World Health Organization (WHO) criteria. Pathological response after surgery, will be based on the proportion of remaining tumor and post-chemotherapy changes, evaluating separately the response in the breast and in the axilla lymph nodes.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to week 12
  Tumor response is defined as the percentage of patients with a complete or partial response out of the patients who had measurable disease at baseline.
Conservative surgery rate | Up to week 15
  To determine the percentage of conservative surgery rate versus other surgery
The Number of Participants Who Experienced Adverse Events (AE) | Through study treatment up to surgery
  According to the Common Terminology Criteria for Adverse Events (CTCAE) version 2.0
Disease-free survival | Up to 5 years since surgery
  Time from the start of treatment to the progression of the disease (if it happens)
Tissue molecular markers and their correlation with response | Up to week 15
  Evaluation of changes in the tumor marker profile before and after treatment in tumor samples obtained before and after chemotherapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Miguel Servet; Study Director, Study Director — Complejo Hospitalrio de Jaén
Locations (10):
- Spain (10):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Complejo Hospitalario Unviesitario A Coruña, A Coruña
  - Hospital Infanta Cristina, Badajoz
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Result] Sanchez-Rovira P, Anton A, Barnadas A, Velasco A, Lomas M, Rodriguez-Pinilla M, Ramirez JL, Ramirez C, Rios MJ, Castella E, Garcia-Andrade C, San Antonio B, Carrasco E, Palacios JL. Classical markers like ER and ki-67, but also survivin and pERK, could be involved in the pathological response to gemcitabine, adriamycin and paclitaxel (GAT) in locally advanced breast cancer patients: results from the GEICAM/2002-01 phase II study. Clin Transl Oncol. 2012 Jun;14(6):430-6. doi: 10.1007/s12094-012-0820-4. PMID 22634531
- See also: Description Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org